CLINICAL TRIAL: NCT00551239
Title: A Randomized Phase III Trial Comparing the Combination of Fludarabine, BBR 2778 (Pixantrone) and Rituximab (FP-R) With the Combination of Fludarabine and Rituximab (F-R) in the Treatment of Patients With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma
Brief Title: Fludarabine and Rituximab With or Without Pixantrone in Treating Patients With Relapsed or Refractory Indolent Non-Hodgkin Lymphoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CTI-CRRI-0807003; CDR0000573364 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-10-22; First posted 2007-10-30 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Leukemia; Lymphoma
Keywords: stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; fludarabine phosphate

ARMS (2):
- Arm I (control) (Active Comparator): Patients receive rituximab IV on day 1 and fludarabine phosphate IV on days 2-4. Treatment repeats every 28 days for up to 6 courses.
  Interventions: Biological: rituximab; Drug: fludarabine phosphate
- Arm II (Experimental): Patients receive rituximab and fludarabine phosphate as in arm I. Patients also receive pixantrone IV on day 2. Treatment repeats every 28 days for up to 6 courses.
  Interventions: Biological: rituximab; Drug: fludarabine phosphate; Drug: pixantrone dimaleate

INTERVENTIONS:
Biological: rituximab — Given IV
Drug: fludarabine phosphate — Given IV
Drug: pixantrone dimaleate — Given IV
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and pixantrone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known whether giving fludarabine together with rituximab is more effective with or without pixantrone in treating indolent non-Hodgkin lymphoma.

PURPOSE: This randomized phase III trial is studying fludarabine and rituximab to compare how well they work with or without pixantrone in treating patients with relapsed or refractory indolent non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the progression-free survival (PFS) of patients with relapsed or refractory indolent non-Hodgkin lymphoma treated with fludarabine phosphate and rituximab with vs without pixantrone.

Secondary

* To compare the overall objective response rate (complete response [CR], unconfirmed complete response [CRu], and partial response [PR]) in these patients.
* To compare the CR and CRu rate in these patients.
* To compare the duration of response and time to progression in these patients.
* To compare the overall survival and disease-specific survival of these patients.
* To compare the safety (including cardiac safety) and tolerability of these regimens in these patients.

OUTLINE: This is a multicenter study. Patients are stratified by Follicular Lymphoma International Prognostic Index (FLIPI) score (0 or 1 vs ≥ 2), number of prior treatments (1 or 2 vs > 2), and prior anti-CD20 regimen (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I (control): Patients receive rituximab IV on day 1 and fludarabine phosphate IV on days 2-4. Treatment repeats every 28 days for up to 6 courses* in the absence of unacceptable toxicity or disease progression.
* Arm II: Patients receive rituximab and fludarabine phosphate as in arm I. Patients also receive pixantrone IV on day 2. Treatment repeats every 28 days for up to 6 courses* in the absence of unacceptable toxicity or disease progression.

NOTE: *Only patients achieving complete response, unconfirmed complete response, or partial response after 4 courses receive courses 5 and 6.

After completion of study therapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed relapsed or refractory indolent non-Hodgkin lymphoma (NHL)

  * Histological assessment must be confirmed by an independent laboratory prior to study randomization

    * Slides from a biopsy or tissue blocks suitable for review must be available
    * Tissue samples may be from the original diagnostic specimen if samples were obtained within the past 24 months, or may be from a biopsy at the time of study entry
    * Re-biopsy must be done prior to study randomization for patients with signs of rapid progression (i.e., lactate dehydrogenase [LDH] level ≥ 2 times upper limit of normal [ULN])
* Any stage disease (with or without B symptoms), including the following:

  * Grade I or II follicular lymphoma, defined as follows:

    * Grade I follicular center cell lymphoma (formerly known as follicular small cleaved)
    * Grade II follicular center cell lymphoma (formerly known as follicular mixed)
  * Small lymphocytic lymphoma or chronic lymphocytic leukemia (CLL)

    * Patients with CLL must have lymph node involvement that is measurable by radiographic techniques
  * Extranodal marginal zone B-cell lymphoma (excluding gastric MALT)
  * Nodal marginal zone B-cell lymphoma (monocytoid B-cell lymphoma)
  * Splenic marginal zone lymphoma (splenic lymphoma with various lymphocytes)
* CD20+ lymphoma (confirmed by immunochemistry)
* Measurable disease

  * At least one objectively bidimensionally measurable lesion as demonstrated by CT scan, spiral CT scan, PET/CT scan, or MRI, that can be followed for response as a target lesion
  * Patients with only skin lesions or only palpable lymph nodes are not eligible
  * Patients with spleen or bone marrow as only site of disease are not eligible
* Patients must have received at least 1 prior therapy

  * Prior treatment with fludarabine phosphate, doxorubicin, and/or mitoxantrone is allowed provided there was a response to treatment (complete response [CR], unconfirmed complete response [CRu], or partial response [PR]) that lasted ≥ 8 months from the start of that therapy
  * Patients refractory to treatments other than anthracycline/anthracenedione, fludarabine phosphate, or rituximab-containing regimens may be eligible for this study
* No HIV-related lymphoma
* No active CNS involvement based on clinical evaluation

  * If the patient requires a diagnostic lumbar puncture due to high risk criteria (i.e., sinus involvement, high LDH, high International Prognostic Index score, or bone marrow involvement), intrathecal chemotherapy (which may include methotrexate, cytarabine, and corticosteroids) may be administered according to institutional standards

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 3 months
* ECOG performance status 0-1
* LVEF ≥ 50% by MUGA scan
* Creatinine ≤ 1.5 times ULN
* Total bilirubin ≤ 1.5 times ULN (CTC grade 1) (patients with Gilbert's syndrome or other hereditary bilirubin defects may be eligible regardless of bilirubin levels)
* AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN if there is hepatic involvement with lymphoma)
* ANC ≥ 1,500/mm³ (≥ 500/mm³ if bone marrow is involved)
* Platelet count ≥ 75,000/mm³ (with no bleeding)
* No known hypersensitivity to the study drugs or to their excipients
* No known type I hypersensitivity or anaphylactic reactions to murine proteins or to any component of rituximab
* No clinically significant cardiovascular abnormalities (i.e., NYHA class III-IV heart disease), including myocardial infarction within the past 6 months, severe arrhythmia, uncontrolled hypertension, or congestive heart failure requiring current active therapy
* No concurrent serious (NCI CTCAE grade 3-4) infection, including infection requiring oral antibiotics or deep-seated or systemic mycotic infections
* No clinical symptoms suggesting unresolved HIV, hepatitis B, or hepatitis C virus infection

  * Patients with seropositivity presumed to be due to prior vaccination against hepatitis B virus or resolved infection are eligible
* No history of another malignancy except curatively treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in remission, or any other cancer from which the patient has been disease-free for 5 years
* No other condition that, in the judgment of the investigator, would place the patient at undue risk, interfere with the results of the study, or make the patient otherwise unsuitable for the study
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after the completion of study treatment

PRIOR CONCURRENT THERAPY:

* Recovered from all acute toxicities from prior therapies (except alopecia or grade 1 peripheral neuropathy)
* No prior treatment with a cumulative dose of doxorubicin equivalent exceeding 450 mg/m²
* More than 4 weeks since prior radiotherapy, chemotherapy, or other therapies for NHL
* More than 5 days since prior systemic corticosteroids for treatment of NHL
* More than 3 months since prior radioimmunotherapy
* More than 4 weeks since prior major thoracic and/or abdominal surgery and recovered
* More than 1 week since prior minor surgery and recovered
* More than 30 days since prior and no other concurrent investigational drugs
* Concurrent corticosteroids (equivalent of 10 mg of prednisone or less per day) allowed provided they are only used to treat concurrent disease (other than NHL)
* No other concurrent systemic anticancer therapy
* No concurrent radiotherapy to target lesions

  * Concurrent palliative radiotherapy to preexisting stable sites of nonmeasurable disease allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Complete response and unconfirmed complete response rate at the end of course 4 and at end of treatment
Overall objective response rate at the end of course 4 and at the end of treatment
Duration of response
Time to progression
Overall survival
Disease-specific survival
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Igor Gorbatchevsky, MD, Study Chair — CTI BioPharma
Locations (1):
- Cell Therapeutics, Incorporated, Seattle, Washington, United States